CLINICAL TRIAL: NCT01335282
Title: Traditional Chinese Medicine Syndrome Identification in Paediatric Neurology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Prof Virginia CN Wong, Department of Peadiatrics and Adolescent Medicine, The University of Hong Kong
Other Study IDs: UW07-163
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Other Diagnoses and Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Traditional Chinese Medicine (TCM) has a history of more than two millenniums. It has been a common practice in China, Taiwan, Japan and Korea and is becoming increasingly popular worldwide in recent decades However, there is no general consensus for treatment of many diseases among TCM practitioners. In some specialties, such as neurology, there is not enough well documented case reports for practitioners to make reference with. Different practitioners may give different opinions according to their own experience and patients often feel frustrated about that.

Therefore, it is worth recording cases of neurological diseases, with accurate western medicine diagnosis and TCM theory explained. Possible TCM treatments can be suggested accordingly. Being an academic research supervised by western medicine doctor, this study can help to suggest more objective opinion with least conflict of interest.

DETAILED DESCRIPTION:
Traditional Chinese Medicine (TCM) has a history of more than two millenniums. It has been a common practice in China, Taiwan, Japan and Korea. In recent decades, it is becoming increasingly popular worldwide(Victor S. Sierpina 2005). Studies in Hong Kong, showed that TCM is quite common among children in Hong Kong, with about a quarter of children consulting a pediatrician are concurrently using Chinese Medicine.(Lee 2006; Li 2006).

However, there is a lack of standardized protocol for treatment of many diseases among TCM practitioners. In some specialties, such as neurology, there is not enough well documented case reports for TCM practitioners to make reference. Different TCM practitioners may give different opinions according to their own experience and patients often feel frustrated about that.

Therefore, it is worth recording cases of neurological diseases, with accurate western medicine diagnosis and TCM theory explained. Possible TCM treatments can be suggested accordingly. Being an academic research supervised by western medicine doctor, this study can help to suggest more objective opinion with least conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving medical care in the Department of Paediatrics and Adolescent Medicine in Queen Mary Hospital or the Duchess of Kent Children's Hospital, and
* Patients (or their care takers) who are able to provide accurate information about their signs and symptoms

Exclusion Criteria:

* Patients (or their care takers) who are unable to report a reliable medical history

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia CN Wong, Professor, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China